CLINICAL TRIAL: NCT02852031
Title: National Pediatric Cardiology Quality Improvement Collaborative (NPC-QIC) - A Collaborative Initiative to Improve Care of Children With Complex Congenital Heart Disease
Brief Title: National Collaborative to Improve Care of Children With Complex Congenital Heart Disease
Acronym: NPC-QIC
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-3866
Record Dates: First submitted 2016-05-19; First posted 2016-08-02 (Estimated); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Hypoplastic Left Heart Syndrome (HLHS)
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypoplastic Left Heart Syndrome: Infants diagnosed with Hypoplastic Left Heart Syndrome (HLHS)
  Interventions: Other: Collaborative Learning Network

INTERVENTIONS:
Other: Collaborative Learning Network

SUMMARY:
The purpose of this initiative is to improve care and outcomes for infants with HLHS by expanding the NPC-QIC national registry to gather clinical care process, outcome, and developmental data on infants with HLHS between diagnosis and 12 months of age, by improving the use of standards into everyday practice across pediatric cardiology centers, and by engaging parents as partners in the process.

DETAILED DESCRIPTION:
The purpose of this initiative is to improve care and outcomes for infants with HLHS by: 1) expanding the established NPC-QIC national registry to gather clinical care process, outcome, and developmental data on infants with HLHS between diagnosis and 12 months of age, 2) improving implementation of consensus standards, tested by teams, into everyday practice across pediatric cardiology centers, and 3) engaging parents as partners in improving care and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Fetuses or newborns diagnosed with HLHS or other univentricular condition
* Intended to undergo Norwood procedure

Exclusion Criteria:

* None

Max Age: 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants diagnosed with HLHS
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-05; Primary Completion 2026-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Relationship between the implementation of changes in care delivery with changes in the process | 15 months
  The purpose of this data sharing is to facilitate QI and research activities. As more information is gathered in this registry, the study team will determine the data analyses methods to determine if the knowledge gained led to changes in care delivery and/or to better patient outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Garick Hill, MD, Principal Investigator — Cininnati Children's Hospital Medical Center
Locations (63):
- United States (61):
  - Children's of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCLA Mattel Children's Hospital, Los Angeles, California
  - Lucile Packard Children's Hospital-Stanford, Palo Alto, California
  - Sutter Medical Center-Sacramento, Sacramento, California
  - UC Davis Children's Hospital, Sacramento, California
  - Rady Children's Hospital, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Cardiac Center, A.I DuPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida-UF Health, Gainesville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Children's Hospital, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Advocate Children's Hospital, Oak Lawn, Illinois
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Ochsner Hospital For Children, Jefferson, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - University of Maryland Children's Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital and Clinics of Minnesota, Minneapolis, Minnesota
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - Batson Children's Hospital-University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital and Medical Center-Omaha, Omaha, Nebraska
  - Cohen Children's Medical Center Northwell Health, New Hyde Park, New York
  - NYU Medical Center, New York, New York
  - Columbia University- NY Presbyterian, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - The Children's Hospital of Montefiore, The Bronx, New York
  - Levine Children's Hospital-Sanger Heart and Vascular Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University Hospitals Case Medical Center - Rainbow Babies & Children's Hospital, Pediatric Heart Center, Cleveland, Ohio
  - Cleveland Clinic Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - PennState Hershey Medical Center--PennState Health Children's Hospital, Harrisburg, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Children's Medical Center of Dallas, Dallas, Texas
  - Cook Childrens Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - UVA Children's Hospital, Charlottesville, Virginia
  - Inova Children's Hospital, Falls Church, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin, American Family Children's, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- The Hospital for Sick Kids- University of Toronto, Toronto, Ontario, Canada
- Evelina London Children's Healthcare, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available.